CLINICAL TRIAL: NCT04372329
Title: A Tailored Sleep Behavior Change Support System to Promote the Use of Continuous Positive Airway Pressure Therapy: Theorizing the Solution
Brief Title: Promoting the Use of CPAP Therapy Among OSA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Alismail (Other)
Responsible Party: Sponsor-Investigator, Sarah Alismail, Principle Investigator, Claremont Graduate University
Organization: Claremont Graduate University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 3726
Record Dates: First submitted 2020-04-25; First posted 2020-05-04 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP4HealthySleep: System 1 (ABAB) (Experimental): Participants in this group will first receive six tailored educational messages per week and weekly feedback messages notifying participants of their CPAP usage on the seventh day for two weeks (type A). Next, they will receive weekly feedback messages only (one message per week) notifying participants of their CPAP usage for two weeks (type B), re-introduction of type A for another two weeks, followed by re-introduction of type B for two weeks.
  Interventions: Behavioral: CPAP4HealthySleep system
- CPAP4HealthySleep: System 2 (BABA) (Experimental): Participants in this group will first receive weekly feedback messages only (one message per week) notifying participants of their CPAP usage for two weeks (type B). Next, they will receive six tailored educational messages per week and weekly feedback messages notifying participants of their CPAP usage on the seventh day for two weeks (type A), re-introduction of type B for another two weeks, followed by re-introduction of type A for two weeks.
  Interventions: Behavioral: CPAP4HealthySleep system

INTERVENTIONS:
Behavioral: CPAP4HealthySleep system — Tailored multimedia messages and tailored feedback messages delivered via web-based system to participants' phones to motivate them to use their CPAP therapy

SUMMARY:
Obstructive sleep apnea (OSA) is the most common sleep breathing disorder in the U.S. Continuous Positive Airway Pressure (CPAP) therapy is the most effective treatment for OSA. However, up to 50% of patients who accept using CPAP therapy fail to adhere to it. This study will evaluate an information systems (IS)-based solution that sends tailored, motivational, educational messages and tailored feedback messages to promote CPAP usage among noncompliant OSA patients. The primary aim of this study is to determine the efficacy of the proposed IS solution and its effect on fostering the use of CPAP therapy among OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of OSA
* Prescribed treatment of CPAP therapy
* Possession of a mobile phone that has multimedia messaging capabilities
* Capacity to consent.

Exclusion Criteria:

* Unable to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in CPAP usage | During 19 weeks
  The average number of hours per week of CPAP usage.
CPAP compliance | 19 weeks
  Compliance of CPAP use characterized by mask-on time at the prescribed pressure for ≥ 4 hours/day for 70% of monitored nights.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Alismail, MS, MPH, Principal Investigator — Claremont Graduate University
Locations (1):
- Pomona Valley Hospital Medical Center Adults and Children Sleep Disorders Center, Claremont, California, United States